CLINICAL TRIAL: NCT03389282
Title: Metabolites of Tear Fluid - Evaluation in a Clinical Pilot Study
Brief Title: Metabolites of Tear Fluid
Acronym: Metabol-T
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Institute of Ophthalmic Research Tuebingen (Unknown); Institute for Clinical Epidemiology and Applied Biometry Tuebingen (Unknown)
Responsible Party: Sponsor
Other Study IDs: AZ 277/2013BO2
Record Dates: First submitted 2017-12-20; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-10

CONDITIONS: Healthy Subjects
Keywords: Tear, Metabolite
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tear fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Tear Sampling — comprehensive eye exam, Schirmer test, break-up time, tear sampling

SUMMARY:
The pilot trial evaluates the use of modified Schirmer strips and is designed to evaluate inter-individual range of metabolites in tear film.

DETAILED DESCRIPTION:
The variability of tear film metabolites should be investigated in a sample of ophthalmologists in preparation for a pilot study in patients eye diseases.

The easy accessibility of the tear fluid and the lack of invasiveness of the study make it promising and sensible to determine the concentration of various tear film metabolites. Because attention has so far focused primarily on the quantitative and qualitative analysis of tear film proteins, many metabolites have so far only been shown to be contained in tears.

However, before the suitability of the measured values as a predictive parameter of the ocular surface for pathologies can be examined and assessed, it is necessary to determine the scattering variables in a sample of healthy volunteers. Thus, reference areas are to be defined for later investigations in order to enable reliable case number planning thereafter.

Repeated determinations at different times and on different days make it possible in particular to detect a time-dependent relationship in view of the dynamic variability of the tear film. The functional significance of certain metabolites can not yet be assessed in the establishment phase. However, the data may provide important information for the interpretation of a later, planned feasibility study with diseased patients or the influence of applied eye drops.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects at age > 18 years

Exclusion Criteria:

* in the case of subjects with a mental disability or legal guardianship, due to possible conflicts for the caregivers, a data evaluation and recording should in principle be dispensed with.
* subjects who have had any eye drops within the last 4 weeks, e.g. lubricants were used
* subjects undergoing clinical examination for symptoms of wetting disorder or morphological changes related to eye disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers without any eye condition and normal anterior surface
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-11-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
concentration of analytes (lipids, proteins/amino acids) | 3 days per patient
  level of analytes (ng/ml)
number of detecatable analytes | 3 days per patient
  number of analytes (lipds, proteins/amino acids)

CONTACTS AND LOCATIONS:
Overall Officials: Focke Ziemssen, MD, Principal Investigator — Center for Ophthalmology, University of Tuebingen
Locations (1):
- University Eye Hospital, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No